CLINICAL TRIAL: NCT05514795
Title: Validity and Reliability of the Thai Version of the Knowledge and Attitudes Survey Regarding Pain (KASRP)
Brief Title: Validity and Reliability of the Thai KASRP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Sasikaan Nimmaanrat, Associate Professor, Prince of Songkla University
Other Study IDs: REC.65-245-8-1
Record Dates: First submitted 2022-08-21; First posted 2022-08-24 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pain is a very common symptom. Pain was found to be a major cause for visiting a doctor. It accounted for 40% of the primary care visits. Pain is also the leading cause of Emergency Department visits. Physicians have a significant role for assessment and management of various kinds of pain.

Knowledge and attitude of doctors (as well as other health care providers) affect their pain management. A survey study using The Knowledge and Attitudes Survey Regarding Pain (KASRP) questionnaire performed in Malaysia revealed that 41.7% of respondents had scores less than 60% regarding pain knowledge. It also revealed that male medical officers had better performance than female medical officers. Anesthesiologist showed the highest mean score. Authors of this study concluded that there is a lack of knowledge and attitude on assessment and management of pain. A similar survey study was performed in Jordan to evaluate health care providers' knowledge and attitudes by using the KASRP. Even doctors had more pain knowledge in comparison to nurses, both of them demonstrated a low level of knowledge and negative attitudes in terms of pain management. A survey study from Iran showed that less than half of health care providers who volunteered to complete a study questionnaire had correct response. Only 9.3% of them thought that they had received sufficient teaching regarding pain and its management.

DETAILED DESCRIPTION:
The Knowledge and Attitudes Survey Regarding Pain (KASRP) The Knowledge and Attitudes Survey Regarding Pain (KASRP) 2014 is a 39-item questionnaire. It comprises of 22 true or false questions and 17 multiple choice questions. Its purpose is to measure knowledge and attitudes of health care providers in regard to pain. It is principally useful as a pre- and post-test measure and can be utilized to rate learning outcomes following educational programs on pain. The KASRP tool was developed in 1987 and has been used extensively since then until present. It has been revised over several years to reflect changes in pain management practice. Its content validity has been established by review of pain specialists. The content of the KASRP tool is derived from standards of pain management such as the American Pain Society (APS), the World Health Organization (WHO), and the National Comprehensive Cancer Network Pain Guidelines. Its construct validity has been established by comparing scores of nurses at various levels of expertise such as students, new graduates, oncology nurses, graduate students, and senior pain experts. The tool was identified as discriminating between levels of expertise. Test-retest reliability was established (r > 0.80) by repeat testing in a continuing education class of nursing staffs (n = 60). Internal consistency reliability was established (alpha r > 0.70) with items reflecting both knowledge and attitude domains.

ELIGIBILITY:
Inclusion Criteria:

* Health care providers

Exclusion Criteria:

* None

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Health care providers
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Validity of the Thai KASRP | Up to 6 months
  Validity of the Thai version of KASRP questionnaire (39 questions, 41 scores)
Reliability of the Thai KASRP | Up to 6 months
  Reliability of the Thai version of KASRP questionnaire (39 questions, 41 scores)

CONTACTS AND LOCATIONS:
Overall Officials: Sasikaan Nimmaanrat, Principal Investigator — Department of Anesthesiology, Faculty of Medicine, Prince of Songkla University
Locations (1):
- Sasikaan Nimmaanrat, Hat Yai, Changwat Songkhla, Thailand